CLINICAL TRIAL: NCT01897987
Title: Follow-up Safety and Efficacy Evaluation on Subjects Who Completed the Initial Stage of PNEUMOSTEM® Phase-II Clinical Trial
Brief Title: Follow-up Safety and Efficacy Evaluation on Subjects Who Completed PNEUMOSTEM® Phase-II Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-CR-009-FU
Record Dates: First submitted 2013-07-04; First posted 2013-07-12 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Human Umbilical Cord Blood Derived Mesenchymal Stem Cells; Bronchopulmonary dysplasia; Premature infants
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pneumostem® (Experimental): A single intratracheal administration of Pneumostem® (1.0 x 10^7 cells/kg)
  Interventions: Biological: Pneumostem®
- normal saline (Placebo Comparator): A single intratracheal administration of normal saline
  Interventions: Biological: normal saline

INTERVENTIONS:
Biological: Pneumostem®
  Other Names: Human umbilical cord blood-derived mesenchymal stem cells
  Arms: Pneumostem®
Biological: normal saline
  Arms: normal saline

SUMMARY:
This is a follow-up study to investigate the long-term safety and efficacy of PNEUMOSTEM® versus placebo, for the treatment of BPD in premature infants. Subjects who participated in and completed the initial stage of the Phase II trial (NCT01828957) will be followed-up until 60 months of corrected age.

DETAILED DESCRIPTION:
Subjects who completed the initial stage of the Phase II clinical trial will be followed-up at 7 additional visits: corrected age of 6, 12,18, 24, 36, 48, and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject who completed the safety and efficacy evaluations in Pneumostem Phase II clinical trial
* Subject with a written consent form signed by a legal representative or a parent upon explanation of the clinical trial

Exclusion Criteria:

* Subject whose parent or legal representative does not agree to participate in the study
* subject who is considered inappropriate to participate in the study by the investigator

Ages: 7 Months to 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Respiratory outcome: readmission rate and duration of the hospital stay due to respiratory infection | 6, 12, 18, 24, 36, 48, and 60 months, corrected age

SECONDARY OUTCOMES:
Whether the subject is receiving medical treatments and if so, duration of the treatment (use of oxygen, steroid, or brochodilator) | 6, 12, 18, 24, 36, 48, and 60 months, corrected age
Number of admissions to Emergency Room | 6, 12, 18, 24, 36, 48, and 60 months, corrected age
  Total number of admissions to Emergency Room and number of admissions to Emergency Room due to resiratory problems
Survival | 6, 12, 18, 24, 36, 48, and 60 months, corrected age
Growth measured by Z-score | 6, 12, 18, 24, 36, 48, and 60 months, corrected age
Neurological developmental status on K-ASQ, Bayley Scale, Gross Motor Function Classification System (GMFCS) for Cerebral Palsy | 24 months, corrected age
Deafness or Blindness | 24 months, corrected age
Number of adverse events | 6, 12, 24,36, 48, and 60 months, corrected age
Significant changes in vital signs | 6, 12, 24, 36, 48, and 60 months, corrected age
Significant changes in physical exam | 6, 12, 24, 36, 48, and 60 months, corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Wonsoon Park, MD, PhD, Principal Investigator — Department of Pediatrics, Samsung Medical Center; Ai-Rhan Kim, MD, PhD, Principal Investigator — Department of Neonatology, Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Ahn SY, Chang YS, Lee MH, Sung S, Kim AR, Park WS. Five-year follow-up of phase II trial of stromal cells for bronchopulmonary dysplasia. Thorax. 2023 Nov;78(11):1105-1110. doi: 10.1136/thorax-2022-219622. Epub 2023 Aug 21. PMID 37604693